CLINICAL TRIAL: NCT00775879
Title: Interest of the Induction With Target-controlled Inhalation of Sevoflurane on Spikes Wave Occurrence
Acronym: SIZE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CHUBX 2004/01
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-05

CONDITIONS: General Anesthesia
Keywords: Général anesthesia; Gynecology
MeSH Terms: interventions — Neoadjuvant Therapy; Sevoflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): 2.5% target concentration
  Interventions: Drug: Induction with Sevoflurane
- B (Active Comparator): 2.5% manually selected
  Interventions: Drug: Induction with Sevoflurane

INTERVENTIONS:
Drug: Induction with Sevoflurane

SUMMARY:
Sevoflurane is widely used for induction of anaesthesia. Several studies showed EEG abnormalities during mask induction with sevoflurane. The aim of our study was to test the induction target concentration of sevoflurane on the spikes wave occurrence.

ELIGIBILITY:
Inclusion Criteria:

* programmed gynecological surgery
* ASA 1 or 2

Exclusion Criteria:

* arterial hypertension
* gastro-oesophageal reflux
* pregnancy
* diabetes
* obesity
* asthma
* tobacco

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2006-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Incidence of spike wave | during anaesthesia induction with sevoflurane

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin JULLIAC, Dr, Principal Investigator — University Hospital, Bordeaux